CLINICAL TRIAL: NCT07403721
Title: A Phase 1/1b Study Evaluating the Safety, Tolerability, and Pharmacokinetics of AMG 436 as Monotherapy and in Combination With Other Therapies in Participants With Microsatellite Instability-high (MSI-H)/Mismatch Repair Deficient (dMMR) Solid Tumors
Brief Title: AMG 436 as Monotherapy and Combination Therapy in Participants With MSI-H/dMMR Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20250004; 2025-524056-63-00 (Other: EU CT Number)
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Metastatic or Locally Advanced Solid Tumors With Microsatellite Instability-high (MSI-H) or Mismatched Repair Deficiency (dMMR)
Keywords: AMG 436; MSI-H; dMMR; Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A (Experimental): AMG 436 monotherapy dose escalation.
  Interventions: Drug: AMG 436
- Part 1B: Food Effect Substudy (Experimental): Participants will receive AMG 436 under fasted and fed conditions (United States only).
  Interventions: Drug: AMG 436
- Part 2 (Experimental): AMG 436 + combination dose escalation.
  Interventions: Drug: AMG 436
- Part 3 (Experimental): AMG 436 monotherapy Dose expansion and optimization.
  Interventions: Drug: AMG 436
- Part 4 (Experimental): AMG 436 + chemotherapy combination dose expansions.
  Interventions: Drug: AMG 436

INTERVENTIONS:
Drug: AMG 436 — AMG 436 will be administered.

SUMMARY:
The primary objectives of this trial are to evaluate the safety profile of AMG 436 and to determine the maximum tolerated dose (MTD) and/or the recommended dose for AMG 436 as monotherapy and in combination with other anti-cancer therapies in participants with MSI-H/dMMR solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (or ≥ legal age within the country if it is older than 18 years).
* Histologically confirmed MSI-H or dMMR metastatic or locally advanced solid tumor by local testing or central testing.
* Tumor tissue (formalin-fixed, paraffin-embedded sample) archival block must be available. Participants without archived tumor tissue may enroll by undergoing tumor biopsy before dosing.
* Disease measurable as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
* Eastern Cooperative Oncology Group performance (ECOG) 0-1.
* Adequate organ function as defined in the protocol.

Exclusion Criteria:

* Participants with primary central nervous system (CNS) tumors.
* Impaired cardiac function or clinically significant cardiac disease.
* Major surgery within 28 days of trial day 1.
* Antitumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, hormonal therapy, or investigational agent) within 21 days of first dose of trial treatment, unless anti-tumor therapy is a therapy with 5 times the half-life being shorter than 21 days (in this case, enrollment may be allowed with washout from prior therapy of < 21 days.
* Radiation therapy within 28 days of the first dose of trial treatment (or local or focal radiotherapy with palliative intent within 14 days of the first dose).
* Gastrointestinal tract disease causing the inability to take per os (PO) medication, malabsorption syndrome, requirement for intravenous (IV) alimentation, uncontrolled inflammatory gastrointestinal disease (eg, Crohn's disease, ulcerative colitis).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2029-04-23 (Estimated); Study Completion 2032-04-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Dose Limiting Toxicity (DLT) | Up to 21 days
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 5 years

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of AMG 436 | Up to 57 days
Minimum Serum Concentration (Cmin) of AMG 436 | Up to 57 days
Area Under the Concentration-time Curve (AUC) Over the Dosing Interval of AMG 436 | Up to 57 days
Time to Achieve Cmax (Tmax) of AMG 436 | Up to 57 days
Part 1B: Cmax of AMG 436 in the Fed and/or Fasted State | Up to 24 days
Part 1B: Tmax of AMG 436 in the Fed and/or Fasted State | Up to 24 days
Part 1B: AUC Over the Dosing Interval of AMG 436 in the Fed and/or Fasted State | Up to 24 days
Confirmed Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 5 years
Duration of Response (DOR) per RECIST v1.1 | Up to 5 years
Time to Response (TTR) per RECIST v1.1 | Up to 5 years
Disease Control Rate (DCR) per RECIST v1.1 | Up to 5 years
Progression-free Survival (PFS) per RECIST v1.1 | Up to 5 years
Overall Survival (OS) per RECIST v1.1 | Up to 5 years
Change From Baseline in Tumor Phosphorylated Checkpoint Kinase 2 (CHK2) Following AMG 436 | Baseline up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this trial will be considered beginning 18 months after the trial has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this trial.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen trial/trials in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com